CLINICAL TRIAL: NCT01882270
Title: Pericoronitis; Oral and Systemic Inflammation
Brief Title: Third Molar Clinical Trials: Pericoronitis Studies
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 05-2846
Record Dates: First submitted 2013-06-17; First posted 2013-06-20 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Pericoronitis
Keywords: pericoronitis; periodontal
MeSH Terms: conditions — Pericoronitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — GCF samples. biofilm samples serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mild Pericoronitis: Those with mild signs/symptoms of pericoronitis affecting at least one lower 3rd molar with adjacent 2nd molar will be monitored for 12 months following study entry or 3 months for those electing to have 3rd molar extraction.

SUMMARY:
The purpose of this research study is to find out if the infection around 3rd molars and the resulting inflammation around the gum also produces a general systemic inflammation.

DETAILED DESCRIPTION:
Relate signs and symptoms of mild pericoronitis, an oral clinical condition characterized by intense inflammation and pain around a lower 3rd molar, to indicators of oral and systemic inflammation in patients seeking treatment for the condition.

ELIGIBILITY:
Inclusion Criteria:

* Mild signs/symptoms of pericoronitis affecting at least one lower 3rd molar with adjacent 2nd molar (spontaneous pain with localized swelling, purulence/drainage) with recommended treatment being removal of 3rd molars,
* Age 18 - 35 years,
* ASA I, II health status,
* AAP 1-3 periodontal status,
* Willingness to participate in the study,
* Geographic proximity to UNC.

Exclusion Criteria:

* Major signs/symptoms of pericoronitis (Temperature >101 , dysphagia, limited mouth opening <20mm incisor, facial swelling/cellulitis, severe uncontrolled discomfort),
* ASA III, IV health status,
* Medical contraindication to full mouth periodontal probing,
* AAP 4 periodontal status,
* Antibiotic treatment within the past 2 months,
* Current tobacco use,
* BMI > 29,
* Pregnancy,
* Non English speaking.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Those with mild signs/symptoms of pericoronitis affecting at least one lower 3rd molar with adjacent 2nd molar with recommended treatment being removal of 3rd molars.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2008-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Quality of Life | one year
  HRQOL data each day for seven days: Subject diary Pain 7pt Likert scale for worst/average pain in past 24h Gracely Scales for current sensory perception/affect Lifestyle, oral function, other symptoms 5pt Likert type scale Global QOL OHIP 14

SECONDARY OUTCOMES:
inflammatory mediators | one year
  For enrolled patients with minor signs and symptoms of pericoronitis:
  1. Assess oral inflammation
     * Levels of "orange/red complex" anaerobic bacteria in biofilm samples from distal of all 2nd molars and distal of affected 3rd molar.
     * Levels of GCF inflammatory mediators, PGE2 and IL-1ß from distal of all 2nd molars and mesial of 1st molars. If the first molar is absent, the mesial of the next most anterior tooth in the quadrant.
  2. Assess the possible association between oral inflammation and systemic inflammation -Serum C-Reactive Protein and IL-6 levels at the time of active symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Ray White, DDS, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC School of Dentistry, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Golden BA, Baldwin C, Sherwood C, Abdelbaky O, Phillips C, Offenbacher S, White RP Jr. Monitoring for periodontal inflammatory disease in the third molar region. J Oral Maxillofac Surg. 2015 Apr;73(4):595-9. doi: 10.1016/j.joms.2014.10.010. Epub 2014 Oct 22. PMID 25544296
- [Derived] Magraw CB, Golden B, Phillips C, Tang DT, Munson J, Nelson BP, White RP Jr. Pain with pericoronitis affects quality of life. J Oral Maxillofac Surg. 2015 Jan;73(1):7-12. doi: 10.1016/j.joms.2014.06.458. Epub 2014 Jul 7. PMID 25262404